CLINICAL TRIAL: NCT02441764
Title: Post-Marketing Surveillance of Halaven Injection in Korean Patients
Brief Title: Halaven Post-Marketing Surveillance (PMS)
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: EKI-PMS-1201
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Halaven; Eribulin Mesylate; locally advanced or metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Halaven: Participants who are prescribed with Halaven per approved prescribing information of Halaven.

SUMMARY:
This is a PMS to observe the safety profile of Halaven in normal clinical practice setting.

ELIGIBILITY:
Participants who are prescribed with Halaven per approved prescribing information of Halaven will be enrolled in the study. This study will be conducted as complete surveillance method; participants who meet the inclusion/exclusion criteria and administrate Halaven for the first time after conclusion of agreement will be enrolled after consent.

Inclusion Criteria:

Participants who meet all of the following criteria will be eligible for inclusion in the study:

1. Participants with following indication: Participants with locally advanced or metastatic breast cancer who have previously received at least two chemotherapeutic regimens which should have included an anthracycline and a taxane.
2. Participants who have verbal or written consent for use of personal and medical information.

Investigators will refer to indications regarding inclusion criteria.

Exclusion Criteria:

1. Hypersensitivity to the active substance or to any of the excipients
2. Breast feeding
3. Pregnancy

Investigators will refer to indications and contraindications regarding exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are prescribed with Halaven per approved prescribing information of Halaven will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Safety of Halaven as a measure of number of participants with adverse events/serious adverse events/adverse drug reactions | Up to 1 year

SECONDARY OUTCOMES:
Tumor response to Halaven treatment | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Busan
  - Chuncheongnam-do
  - Chungcheongbuk-do
  - Chungcheongnam-do
  - Daegu
  - Gwangju
  - Gyeonggi-do
  - Gyeongsanbuk-do
  - Gyeongsannam-do
  - Jeollabuk-do
  - Jeollanam-do
  - Seoul